CLINICAL TRIAL: NCT01225549
Title: A Double-blind, Double-dummy, Randomised, Placebo-controlled, 4-way, Crossover, Multi-centre Phase II Study With Budesonide as an Active Control to Evaluate the Efficacy and Safety of 2 Doses of Inhaled AZD5423 Over 7 Days in Patients With Mild Allergic Asthma Challenged With an Inhaled Allergen
Brief Title: The Study Will Evaluate the Efficacy of AZD5423 in Patients With Mild Asthma Challenged With an Inhaled Allergen
Acronym: Allergen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D2340C00005
Record Dates: First submitted 2010-10-15; First posted 2010-10-21 (Estimated); Results first posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Asthma
Keywords: Allergen Challenge; Asthma; Inhaled selective glucocorticoid receptor agonist (iSEGRA)
MeSH Terms: conditions — Asthma | interventions — 2,2,2-trifluoro-N-(1-((1-(4-fluorophenyl)-1H-indazol-5-yl)oxy)-1-(3-methoxyphenyl)-2-propanyl)acetamide; Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental): AZD5423 75ug
  Interventions: Drug: AZD5423; Drug: Placebo
- 2 (Experimental): AZD5423 300ug
  Interventions: Drug: AZD5423; Drug: Placebo
- 3 (Active Comparator): Budesonide 200 microgram
  Interventions: Drug: Budesonide 200 microgram; Drug: Placebo
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5423 — Suspension for nebulisation once daily 7 days
  Arms: 1; 2
Drug: Budesonide 200 microgram — Dry powder for inhalation twice daily 7 days
  Other Names: Pulmicort
  Arms: 3
Drug: Placebo — Solution for nebulisation once daily 7 days
  Arms: 3; 4
Drug: Placebo — Solution for nebulisation once daily 7 days
  Arms: 1; 2; 4

SUMMARY:
The purpose of this study is to evaluate the efficacy of AZD5423 in patients with mild asthma challenged with an inhaled allergen.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age
* Pre-bronchodilatory FEV1 ≥70% of predicted normal allergic asthmatic with a history of episodic wheeze
* Positive allergen induced early and late airway bronchoconstriction showing ≥ 20% fall in FEV1 for the early and ≥ 15% for the late response
* Positive skin prick test to common aeroallergens

Exclusion Criteria:

* Any clinically significant disease or disorder
* Any clinically relevant abnormal finding at screening examinations
* Smoker or ex-smoker who has stopped smoking < 12 months prior to study start
* Worsening of asthma or respiratory infection within 6 weeks from visit 1
* Allergen-specific immunotherapy within 6 months prior to visit 1

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christer Hultquist, Study Director — AstraZeneca R&D, Mölndal, Sweden
Locations (4):
- Canada (4):
  - Research Site, Calgary, Alberta
  - Research Site, Hamilton, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Gauvreau GM, Boulet LP, Leigh R, Cockcroft DW, Killian KJ, Davis BE, Deschesnes F, Watson RM, Swystun V, Mardh CK, Wessman P, Jorup C, Aurivillius M, O'Byrne PM. A nonsteroidal glucocorticoid receptor agonist inhibits allergen-induced late asthmatic responses. Am J Respir Crit Care Med. 2015 Jan 15;191(2):161-7. doi: 10.1164/rccm.201404-0623OC. PMID 25473939
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=203&filename=D2340C00005.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from 4 centres in the AllerGen CIC group in Canada.
Pre-assignment Details: Total 27 patients enrolled, 20 (74.1%) patients were randomised to receive a treatment sequence consisting of 4 different treatment in random order. From 20 randomised patients, 18 (90%) patients completed the study and 2 (10%) patients were withdrawn from the study due to consumption of disallowed medication
Groups:
- ACBP: AZD5423 75 µg followed by budesonide 200 µg bid followed by AZD5423 300 µg od followed by placebo
- APBC: AZD5423 75 µg followed by placebo followed by AZD5423 300 µg od followed by budesonide 200 µg bid
- BACP: AZD5423 300 µg od followed by AZD5423 75 µg followed by budesonide 200 µg bid followed by placebo
- BPCA: AZD5423 300 µg od followed by placebo followed by budesonide 200 µg bid followed by AZD5423 75 µg
- CAPB: Budesonide 200 µg bid followed by AZD5423 75 µg followed by placebo followed by AZD5423 300 µg od
- CBAP: Budesonide 200 µg bid followed by AZD5423 300 µg od followed by AZD5423 75 µg followed by placebo
- CBPA: Budesonide 200 µg bid followed by AZD5423 300 µg od followed by placebo followed by AZD5423 75 µg
- PBAC: Placebo followed by AZD5423 300 µg od followed by AZD5423 75 µg followed by budesonide 200 µg bid
- PCAB: Placebo followed by budesonide 200 µg bid followed by AZD5423 75 µg followed by AZD5423 300 µg od
- PCBA: Placebo followed by budesonide 200 µg bid followed by AZD5423 300 µg od followed by AZD5423 75 µg
Period: Period 1 - First Treatment Period
Arm/Group | ACBP | APBC | BACP | BPCA | CAPB | CBAP | CBPA | PBAC | PCAB | PCBA
Started | 1 | 4 | 3 | 1 | 1 | 1 | 3 | 1 | 4 | 1
Completed | 1 | 4 | 3 | 1 | 1 | 1 | 3 | 1 | 4 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 - Washout
Arm/Group | ACBP | APBC | BACP | BPCA | CAPB | CBAP | CBPA | PBAC | PCAB | PCBA
Started | 1 | 4 | 3 | 1 | 1 | 1 | 3 | 1 | 4 | 1
Completed | 1 | 4 | 3 | 1 | 1 | 1 | 3 | 1 | 4 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3 - Second Treatment Period
Arm/Group | ACBP | APBC | BACP | BPCA | CAPB | CBAP | CBPA | PBAC | PCAB | PCBA
Started | 1 | 4 | 3 | 1 | 1 | 1 | 3 | 1 | 4 | 1
Completed | 1 | 4 | 3 | 1 | 1 | 1 | 3 | 1 | 4 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4 - Washout
Arm/Group | ACBP | APBC | BACP | BPCA | CAPB | CBAP | CBPA | PBAC | PCAB | PCBA
Started | 1 | 4 | 3 | 1 | 1 | 1 | 3 | 1 | 4 | 1
Completed | 1 | 3 | 3 | 1 | 1 | 1 | 3 | 1 | 4 | 1
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disallowed medication | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 5 - Third Treatment Period
Arm/Group | ACBP | APBC | BACP | BPCA | CAPB | CBAP | CBPA | PBAC | PCAB | PCBA
Started | 1 | 3 | 3 | 1 | 1 | 1 | 3 | 1 | 4 | 1
Completed | 1 | 3 | 3 | 1 | 1 | 1 | 3 | 1 | 4 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 6 - Washout
Arm/Group | ACBP | APBC | BACP | BPCA | CAPB | CBAP | CBPA | PBAC | PCAB | PCBA
Started | 1 | 3 | 3 | 1 | 1 | 1 | 3 | 1 | 4 | 1
Completed | 1 | 3 | 3 | 0 | 1 | 1 | 3 | 1 | 4 | 1
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disallowed medication | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 7 - Fourth Treatment Period
Arm/Group | ACBP | APBC | BACP | BPCA | CAPB | CBAP | CBPA | PBAC | PCAB | PCBA
Started | 1 | 3 | 3 | 0 | 1 | 1 | 3 | 1 | 4 | 1
Completed | 1 | 3 | 3 | 0 | 1 | 1 | 3 | 1 | 4 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Baseline Total: Total number of patients randomised and treated in the study
Arm/Group | Baseline Total
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: Years] | 29.6 [18 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 19
  Others | 1

OUTCOME MEASURES:

1. Primary Outcome: Late Allergic Response (LAR) by Assessment of Minimum Percentage of FEV1 3-7 Hours Post Allergen Challenge Compared to Pre Allergen Challenge FEV1
Description: LAR was assessed on Day 6 as minimum percentage of FEV1 over 3 to 7 hours based on the analysis of the minimum percentage of FEV1 remaining over 3 to 7 hours post allergen challenge (post AC) compared to pre allergen challenge (pre AC) FEV1
Time Frame: From Randomization to end of treatment
Population: PD Analysis set
Measure: Geometric Mean (Full Range); unit: Percentage
Groups:
- Arm 1 - 75ug AZD5423: 75ug AZD5423 administered once daily in any of the first, second, third or fourth period of a particular sequence.
- Arm 2 - 300ug AZD5423: 300ug AZD5423 administered once daily in any of the first, second, third or fourth period of a particular sequence.
- Arm 3 - 2x200ug Budesonide: 200µg budesonide administered twice daily in any of the first, second, third or fourth period of a particular sequence.
- Arm 4 - Placebo: Placebo administered in any of the first, second, third or fourth period of a particular sequence.
Arm/Group | Arm 1 - 75ug AZD5423 | Arm 2 - 300ug AZD5423 | Arm 3 - 2x200ug Budesonide | Arm 4 - Placebo
Number analyzed (Participants) | 19 | 19 | 19 | 19
Percentage | 90.97 [73.20 to 100.00] | 91.32 [76.80 to 101.60] | 87.28 [56.60 to 103.20] | 85.83 [69.60 to 102.80]

2. Secondary Outcome: Early Allergic Response (EAR) by Assessment of Minimum Percentage of FEV1 0-3 h Post Allergen Challenge
Description: Minimum Percentage of FEV1 over 0 to 3 hours post allergen challenge compared to pre allergen challenge FEV1
Time Frame: From Randomization to end of treatment
Population: PD Analysis set
Measure: Geometric Mean (Full Range); unit: Percentage
Arm/Group | Arm 1 - 75ug AZD5423 | Arm 2 - 300ug AZD5423 | Arm 3 - 2x200ug Budesonide | Arm 4 - Placebo
Number analyzed (Participants) | 19 | 19 | 19 | 19
Percentage | 69.75 [41.00 to 94.00] | 69.57 [41.80 to 92.60] | 67.98 [41.60 to 92.40] | 69.30 [35.20 to 92.60]

3. Secondary Outcome: Area Under the Curve (AUC) for FEV1 Over 0-3 and 3-7 h Post Allergen Challenge
Description: AUC was assessed as average percentage of FEV1 remaining 0 to 3 hours and 3 to 7 hours post allergen challenge compared to pre allergen challenge FEV1
Time Frame: From Randomization to end of treatment
Population: PD Analysis set
Measure: Geometric Mean (Full Range); unit: Percentage
Arm/Group | Arm 1 - 75ug AZD5423 | Arm 2 - 300ug AZD5423 | Arm 3 - 2x200ug Budesonide | Arm 4 - Placebo
Number analyzed (Participants) | 19 | 19 | 19 | 19
Percentage
  AUC over 0-3 (Average EAR) | 83.82 [64.10 to 95.25] | 83.71 [65.70 to 96.68] | 81.90 [56.50 to 93.90] | 82.26 [57.10 to 97.97]
  AUC over 3-7 (Average LAR) | 96.30 [87.62 to 104.67] | 96.53 [85.70 to 103.93] | 93.39 [69.69 to 107.34] | 92.50 [80.77 to 106.23]

4. Secondary Outcome: Airway Hyperresponsiveness by Assessment of Methacholine PC20
Description: The methacholine challenge was performed on Day 1 (pre dose), Day 5 ([post dose] pre AC), and Day 7 ([post dose] 24 hours post AC)
Time Frame: Day 1 (pre-dose)
Population: PD Analysis set
Measure: Geometric Mean (Full Range); unit: mg/mL
Arm/Group | Arm 1 - 75ug AZD5423 | Arm 2 - 300ug AZD5423 | Arm 3 - 2x200ug Budesonide | Arm 4 - Placebo
Number analyzed (Participants) | 19 | 19 | 19 | 20
mg/mL | 1.560 [0.11 to 32.00] | 1.651 [0.14 to 36.80] | 1.688 [0.08 to 17.75] | 1.538 [0.07 to 53.70]

5. Secondary Outcome: Airway Hyperresponsiveness by Assessment of Methacholine PC20
Description: as for outcome 4
Time Frame: Day 5 ([post-dose] pre allergen challenge)
Measure: Geometric Mean (Full Range); unit: mg/mL
Arm/Group | Arm 1 - 75ug AZD5423 | Arm 2 - 300ug AZD5423 | Arm 3 - 2x200ug Budesonide | Arm 4 - Placebo
Number analyzed (Participants) | 19 | 19 | 19 | 20
mg/mL | 1.755 [0.13 to 32.00] | 2.693 [0.26 to 64.00] | 2.477 [0.19 to 18.70] | 2.034 [0.09 to 53.80]

6. Secondary Outcome: Airway Hyperresponsiveness by Assessment of Methacholine PC20
Description: as for outcome 4
Time Frame: Day 7 ([post-dose] 24 hours post allergen challenge)
Measure: Geometric Mean (Full Range); unit: mg/mL
Arm/Group | Arm 1 - 75ug AZD5423 | Arm 2 - 300ug AZD5423 | Arm 3 - 2x200ug Budesonide | Arm 4 - Placebo
Number analyzed (Participants) | 17 | 19 | 19 | 18
mg/mL | 2.017 [0.21 to 32.00] | 2.007 [0.15 to 45.89] | 1.666 [0.06 to 17.19] | 1.214 [0.06 to 35.10]

7. Secondary Outcome: Changes in Sputum Eosinophils Differentials (Percentage)
Description: The change form baseline in percentage of sputum eosinophils was assessed on Day 5 (post dose) ,Day 6 ([post dose] 7 hours post allergen challenge) and Day 7 ([post dose] 24 hours post allergen challenge)
Time Frame: Day 5 (post dose)
Population: PD Analysis set
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Arm 1 - 75ug AZD5423 | Arm 2 - 300ug AZD5423 | Arm 3 - 2x200ug Budesonide | Arm 4 - Placebo
Number analyzed (Participants) | 16 | 15 | 15 | 16
Percentage | 1.891 (8.375) | -3.2 (9.162) | -1.825 (4.342) | -0.016 (1.835)

8. Secondary Outcome: Changes in Sputum Eosinophils Differentials (Percentage)
Description: as for outcome 7
Time Frame: Day 6 ([post dose] 7 hours post allergen challenge)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Arm 1 - 75ug AZD5423 | Arm 2 - 300ug AZD5423 | Arm 3 - 2x200ug Budesonide | Arm 4 - Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 15
Percentage | 0.633 (6.011) | 0.592 (9.658) | 7.500 (11.800) | 12.333 (14.260)

9. Secondary Outcome: Changes in Sputum Eosinophils Differentials (Percentage)
Description: as for outcome 7
Time Frame: Day 7 ([post dose] 24 hours post allergen challenge)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Arm 1 - 75ug AZD5423 | Arm 2 - 300ug AZD5423 | Arm 3 - 2x200ug Budesonide | Arm 4 - Placebo
Number analyzed (Participants) | 16 | 14 | 15 | 14
Percentage | 0.688 (8.230) | 2.286 (15.417) | 6.967 (11.697) | 5.634 (5.520)

ADVERSE EVENTS:
Groups:
- Arm 3 - 2x200ug Budesonide: 2x200ug budesonide administered twice daily in any of the first, second, third or fourth period of a particular sequence.
Arm/Group | Arm 1 - 75ug AZD5423 | Arm 2 - 300ug AZD5423 | Arm 3 - 2x200ug Budesonide | Arm 4 - Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 8/19 | 1/19 | 9/19 | 9/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - 75ug AZD5423 (N=19) | Arm 2 - 300ug AZD5423 (N=19) | Arm 3 - 2x200ug Budesonide (N=19) | Arm 4 - Placebo (N=20)
CONJUNCTIVITIS (Eye disorders) | 0 | 0 | 0 | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0 | 0 | 0
DRY MOUTH (Gastrointestinal disorders) | 1 | 0 | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 1 | 0 | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0 | 0 | 0
PYREXIA (General disorders) | 0 | 0 | 1 | 0
BRONCHITIS (Infections and infestations) | 0 | 0 | 2 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 0 | 1 | 0
PHARYNGITIS BACTERIAL (Infections and infestations) | 0 | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 0
VIRAL PHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
SCRATCH (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
HELICOBACTER TEST POSITIVE (Investigations) | 0 | 1 | 0 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
HEADACHE (Nervous system disorders) | 2 | 0 | 1 | 1
INSOMNIA (Psychiatric disorders) | 0 | 0 | 1 | 0
DYSMENORRHOEA (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 2
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Of the 27 patients enrolled, 20 (74.1%) patient were randomised to receive a treatment sequence consisting of 4 different treatment in random order. 19 patients completed each individual treatment period and 17 patients completed all 4 treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall not publish any results until (i) the date of the first Study results publication, or in case of a Multi-Centre Study the first Multi-Centre Results publication, agreed by the participating sites, and (ii) the end of the eighteen (18) month period following the completion or early termination of the Study at all participating sites.